CLINICAL TRIAL: NCT02677090
Title: Fiber Tolerability In Children Aged 3-7 Year
Acronym: Fiber - TIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 15.10.NRC
Record Dates: First submitted 2016-01-29; First posted 2016-02-09 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-01

CONDITIONS: Signs and Symptoms, Digestive
Keywords: Fiber tolerability; Children
MeSH Terms: conditions — Signs and Symptoms, Digestive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo (including Maltodextrin)
- Dose 1 - Promitor® (Active Comparator): Investigational product Dose 1
  Interventions: Drug: Dose 1 - Promitor®
- Dose 2 - Promitor® (Active Comparator): Investigational product Dose 2
  Interventions: Drug: Dose 2 - Promitor®
- Dose 3 - Promitor® (Active Comparator): Investigational product Dose 3
  Interventions: Drug: Dose 3 - Promitor®

INTERVENTIONS:
Drug: Placebo (including Maltodextrin)
  Arms: Placebo
Drug: Dose 1 - Promitor®
  Arms: Dose 1 - Promitor®
Drug: Dose 2 - Promitor®
  Arms: Dose 2 - Promitor®
Drug: Dose 3 - Promitor®
  Arms: Dose 3 - Promitor®

SUMMARY:
Determination of the digestive tolerability of the PROMITOR® in children from 3 to 7 years old.

DETAILED DESCRIPTION:
The aim of the trial is to determine, using a dose escalation design, the digestive tolerability of the PROMITOR®given at the doses of 6, then 9 and finally 12 g (corresponding to 4, 6, and 8 g of fibers respectively) twice a day with the meals of the morning and of the evening versus control (maltodextrin, no fiber) over one week of intake in children from 3 to 7 years old.

As it is an exploratory study there is no categorization between primary and secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children
2. Aged between 3 and 7 years old
3. Acceptance of the taste of the product
4. Having breakfast on daily basis
5. Consent and/or assent received according to regulation
6. Informed consent of both parents/guardians (in respect with the French regulation)
7. Parents/guardians affiliated to a health insurance (in respect with the French regulation)

Exclusion Criteria:

1. Specific food regimen
2. Intolerability or food allergy
3. Antibiotic or any medication impacting the gut transit during the 2 weeks before the study
4. Chronic gastrointestinal disease
5. Gastroenteritis in the 2 weeks preceding the study
6. Constipation or diarrhea based on ROMEIII criteria (in average: more than 3 stools per day or less than 3 stools per week)
7. Children and parents expected not to understand and perform the trial correctly (i.e.: troubles in learning and/or speaking)
8. Child in a situation which, in the opinion of the principal investigator, could interfere with the optimal participation to the study or constitute a particular risk of non-compliance
9. Having participated in another clinical trial for 1 month, or currently participating in a clinical trial
10. Under legal protection or deprived from his rights following administrative or judicial decision (in respect with the French regulation)

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the digestive tolerability of the Investigational Product (abdominal pain) using analog visual scale | 7 days of intake
  Using analog visual scale
Assessment of the digestive tolerability of the Investigational Product (rumbling) using analog visual scale | 7 days of intake
  Using analog visual scale
Assessment of the digestive tolerability of the Investigational Product (bloating) using analog visual scale | 7 days of intake
  Using analog visual scale
Assessment of the digestive tolerability of the Investigational Product (flatulence) using analog visual scale | 7 days of intake
  Using analog visual scale
Assessment of the digestive tolerability of the Investigational Product (stools consistency & frequency) using analog visual scale | 7 days of intake
  Using analog visual scale

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No